CLINICAL TRIAL: NCT05821114
Title: The Effects of High-Flow Nasal Cannula and Body Position On Atelectasis Using Electric Impedance Tomography in Children Awakening From Propofol Anesthesia: A Pilot Randomized Controlled Trial.
Brief Title: End-Expiratory Lung Volume in Children Awakening From Propofol Anesthesia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Hee-Soo Kim, professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2302-129-1408
Record Dates: First submitted 2023-04-07; First posted 2023-04-20 (Actual); Last update posted 2023-04-20 (Actual); Status verified 2023-04

CONDITIONS: Atelectasis, Postoperative Pulmonary
MeSH Terms: conditions — Pulmonary Atelectasis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- high flow oxygen (Experimental): Oxygen supply (2L/kg/min.) during awakening from propofol anesthesia
  Interventions: Other: Head elevation_H; Other: Supine_H
- Low flow oxygen (Active Comparator): Oxygen supply (0.3L/kg/min.) during awakening from propofol anesthesia
  Interventions: Other: Head elevation_L; Other: Supine_L

INTERVENTIONS:
Other: Head elevation_H — High flow_Head-elevation
  Arms: high flow oxygen
Other: Supine_H — High flow_Supine
  Arms: high flow oxygen
Other: Head elevation_L — Low flow_head elevation
  Arms: Low flow oxygen
Other: Supine_L — Low flow_supine
  Arms: Low flow oxygen

SUMMARY:
The goal of this pilot randomized clinical trial is to test the effects of high flow nasal oxygen and head elevation during awakening from propofol anesthesia in pediatric patients undergoing airway surgery.

The main question[s] it aims to answer are:

* High flow oxygen can decrease the occurence of atelectasis during awakening from propofol anesthesia in pediatric patients?
* Head elevation can decrease the occurence of atelectasis during awakening from propofol anesthesia in pediatric patients?

Researchers will compare high flow oxygen vs low flow oxygen group to see if the use of high flow oxygen decrease the occurence of atelectasis during awakening from propofol anesthesia.

And in each group, the patients will be assigned to supine position vs head elevation position to compare the effects of head elevation during awakening from propofol anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients undergoing airway surgery with high flow nasal oxygen

Exclusion Criteria:

* Loss of spontaneous ventilation during surgery
* less than 1 months
* cyanotic patients

Ages: 1 Month to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 52 (Estimated)
Dates: Start 2023-04-07 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in Electric Impedance Tomography parameter | from induction of anesthesia to end of operation, about 3 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Hee-Soo Kim, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided